CLINICAL TRIAL: NCT00504595
Title: A 12-week, Phase II, Multi-center, Randomized, Double-blind, Placebo-controlled Study to Assess the Response to Treatment (ACR20) and to Determine a Biomarker Profile in Adult Patients With Established Rheumatoid Arthritis Responding to ACZ885 (Anti-interleukin-1beta Monoclonal Antibody) as Compared to Healthy Subjects Exposed to ACZ885
Brief Title: Safety and Efficacy of ACZ885 in Adult Patients With Established Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CACZ885A2207
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Results first posted 2011-06-23 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACZ885 (Experimental): Healthy Volunteers: Single administration of 600 mg of ACZ885 (Canakinumab) Intravenous (IV) on Day 1.
  Rheumatoid Arthritis (RA) Patients: Dose of 600 mg of ACZ885 (Canakinumab) Intravenous (IV) on Day 1, Day 15, and Day 43.
  Interventions: Drug: ACZ885 (investigational)
- Placebo (Placebo Comparator): Healthy Volunteers: Single administration of 600 mg of Placebo Intravenous (IV) on Day 1.
  Rheumatoid Arthritis (RA) Patients: Dose of 600 mg of Placebo Intravenous (IV) on Day 1, Day 15, and Day 43.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACZ885 (investigational) — The ACZ885 was supplied in 6 mL colorless glass vials each containing nominally 150 mg ACZ885 (with 20% overfill). The vials were kept at 2-8°C. At the investigator's site, solutions for infusion were prepared depending on the volume and dose administered.
  Other Names: Canakinumab
  Arms: ACZ885
Drug: Placebo — Matching placebo of ACZ885 was supplied in the form of a lyophilized cake (Powder for Solution for Infusion). At the investigator's site, solutions for infusion were prepared depending on the volume and dose administered.
  Arms: Placebo

SUMMARY:
This study was intended to assess the safety, efficacy, and response to treatment using the American College of Rheumatology (ACR) criteria of 20% improvement in symptoms (ACR20) and to investigate a potential biomarker profile in adult patients with established rheumatoid arthritis

ELIGIBILITY:
Inclusion Criteria:

RA patients:

* Male and female patients aged 18 - 75 years (inclusive).
* Body weight between 50 and 100 kg (inclusive).
* Post menopausal or surgically sterile female patients are allowed. Female patients of child-bearing potential may participate if they are already on a stable dose of methotrexate. Additional birth control details to be provided at screening. Male patients must use an effective contraception method during the study and at least for 2 months following the completion/discontinuation of the study.
* Diagnosis of RA, classified by American Rheumatism Association 1987 revised criteria. Disease duration of at least 6 months is essential.
* Functional status class I, II or III classified according to the American College of Rheumatology 1991 revised criteria.
* Active disease evaluation (≥ 6 tender and ≥ 6 swollen joints)
* Prior treatment with 1-3 disease-modifying anti-rheumatic drugs (DMARDs) - Patients should have failed at least 1 DMARD but should not be deemed "refractory to all therapies". It is expected that patients are on a current treatment with methotrexate ≤ 25 mg/week and with the current dose stable for at least 3 months, however patients who did not tolerate MTX may also be considered. All patients will take folic acid 1 mg daily, or 5 mg weekly post MTX dose, to minimize toxicity, according to local guidelines. In addition to methotrexate, patients may be on either a stable dose of non-steroidal anti-inflammatory drugs (NSAIDs) and/or a stable dose of oral corticosteroids (prednisone or equivalent ≤ 10 mg daily) for at least 4 weeks prior to randomization. Patients who failed any DMARDs will be allowed.
* Negative purified protein derivative (PPD) tuberculin skin test reaction (PPD 5 tuberculin units or as according to local standard practice).

Exclusion Criteria:

RA patients:

* Previous treatment with anti-Tumor Necrosis Factor (TNF)-α or anti IL-1 therapy (or other biological therapy), immunosuppressive agents such as cyclosporine, mycophenolate or tacrolimus. The following washout period will be required for such patients to be eligible to participate in the trial.

  1. 2 months washout prior to screening for etanercept or adalimumab
  2. 3 months washout prior to screening for infliximab
  3. 3 months washout prior to screening for rituximab
  4. 1 month washout prior to screening for cyclosporine, mycophenolate and tacrolimus.
* If patient has been discontinued from other DMARDs (disease modifying antirheumatic drugs) for lack of efficacy or toxicity, the patient should be at least 1 month off the agent.
* Patients with congestive heart failure, QT prolongation syndrome or poorly controlled diabetes mellitus. Patients with a history of QTc prolongation will be excluded.
* Patients who have received intra-articular or systemic corticosteroid injections having been required for treatment of acute RA flare (not being part of a regular therapeutic regimen) within 4 weeks prior to randomization.
* Exclusion criteria 2-6 of the Health Volunteer section also applies here.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (4):
- Novartis Investigative site, Moscow, Russia
- Novartis investigative site, Barcelona, Spain
- Novartis Investigative site, Bern, Switzerland
- Novartis investigative site, Istanbul, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Groups:
- ACZ885 (Canakinumab) : RA Patients: Patients with Rheumatoid Arthritis RA taking 600 mg of ACZ885 (Canakinumab) Intravenous (IV) on Day 1, Day 15, and Day 43.
- ACZ885 (Canakinumab) : Healthy Volunteers: Healthy Volunteers taking 600 mg of ACZ885 (Canakinumab) Intravenous (IV) on Day 1
- Placebo Comparator: RA Patients: Rheumatoid Arthritis patients who received placebo Intravenous (IV) on Day 1, Day 15 and Day 43.
- Placebo Comparator: Healthy Volunteers: Healthy Volunteers who received placebo Intravenous (IV) at Day 1.
Period: Overall Study
Arm/Group | ACZ885 (Canakinumab) : RA Patients | ACZ885 (Canakinumab) : Healthy Volunteers | Placebo Comparator: RA Patients | Placebo Comparator: Healthy Volunteers
Started | 50 | 10 | 10 | 10
Completed | 49 | 10 | 8 | 10
Not Completed | 1 | 0 | 2 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACZ885 (Canakinumab) : RA Patients | ACZ885 (Canakinumab) : Healthy Volunteers | Placebo Comparator: RA Patients | Placebo Comparator: Healthy Volunteers | Total
Number analyzed (Participants) | 50 | 10 | 10 | 10 | 80
Age Continuous [Mean (Standard Deviation); unit: Years] | 54.4 (13.42) | 28.8 (7.42) | 46.2 (12.83) | 28.0 (5.52) | 46.9 (16.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 4 | 9 | 2 | 57
  Male | 8 | 6 | 1 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Response to Treatment (ACR20) in Adult Patients With Established Rheumatoid Arthritis (RA)
Description: At each post-dose visit, an ACR20 responder was defined as someone who achieved at least 20% improvement in the tender and the swollen 28-joint count, and 20% improvement in at least 3 of the following 5 measures::
  * Patient's pain assessment (Visual Analogue Scale (VAS) 100 mm)
  * Patient's global assessment of disease activity (VAS 100 mm)
  * Physician's global assessment of disease activity (VAS 100 mm)
  * Patient self-assessed disability (Health Assessment Questionnaire (HAQ) score)
  * Acute phase reactant (high sensitivity C-reactive Protein (hsCRP))
Time Frame: 6 weeks and 12 weeks
Population: The Safety Analysis Set consisted of all subjects who received at least one dose of study medication. The analysis used last observation carried forward (LOCF) imputation for missing values.
Measure: Number; unit: Participants
Arm/Group | ACZ885 (Canakinumab) : RA Patients | Placebo Comparator: RA Patients
Number analyzed (Participants) | 50 | 10
Participants
  ACR20 response rate at 6 weeks | 17 | 2
  ACR20 response rate at 12 weeks | 27 | 2

2. Secondary Outcome: Efficacy of ACZ885 by Assessing the Response to Treatment Using the Simple Disease Index (SDAI)
Description: SDAI is derived by the number of swollen joints and tender joints using the 28-joint count (tender28 and swollen28). SDAI measures the high sensitivity C-reactive protein (hsCRP) level, patient's global disease activity (PGDA) and evaluator's global disease activity (EGDA). PGDA and EGDA are measured on a 100 mm Visual Analogue Scale (VAS), ranging from no arthritis activity to maximal arthritis activity. SDAI = tender28 + swollen28 + CRP + (PGDA/10) + (EGDA/10). Lower scores indicate less disease activity.
Time Frame: 6 weeks and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- ACZ885 (Canakinumab): RA Patients: Patients with Rheumatoid Arthritis (RA) taking 600 mg of ACZ885 (Canakinumab) Intravenous (IV) on Day 1, Day 15, and Day 43.
- Placebo Comparator: RA Patients: Patients with Rheumatoid Arthritis (RA) who received placebo Intravenous (IV) on Day 1, Day 15 and Day 43.
Arm/Group | ACZ885 (Canakinumab): RA Patients | Placebo Comparator: RA Patients
Number analyzed (Participants) | 50 | 10
Scores on a scale
  6 Weeks | 32.623 (13.6218) [-1.04 to 0.17] | 33.841 (15.0053) [-10.75 to 4.83]
  12 Weeks | 29.163 (13.0927) [-1.38 to -0.01] | 32.412 (12.2633) [-12.41 to 2.89]

3. Secondary Outcome: Efficacy of ACZ885 (Canakinumab) by Assessing the Response to Treatment Using the Disease Activity Score (DAS28)
Description: DAS28 is derived by the number of swollen joints and tender joints using the 28-joint count (tender28 and swollen28). DAS28 measures the C-reactive protein (CRP) (in mg/L) and the patient's general health (GH). GH is measured on a 100 mm Visual Analogue Scale (VAS), ranging from no arthritis activity to maximal arthritis activity. DAS28 = 0.56*√(tender28) + 0.28*√(swollen28) + 0.36*log_e(CRP+1) + 0.014*PGDA + 0.96. Lower scores indicate less disease activity.
Time Frame: 6 weeks and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ACZ885 (Canakinumab) : RA Patients | Placebo Comparator: RA Patients
Number analyzed (Participants) | 50 | 10
Scores on a scale
  6 Weeks | 5.088 (1.1148) | 5.397 (1.0591)
  12 Weeks | 4.853 (1.1879) | 5.400 (0.9321)

ADVERSE EVENTS:
Time Frame: 18 Weeks (12 Week treatment period + 6 Week Follow-up period)
Groups:
- ACZ885 (Canakinumab): Healthy Volunteers: Healthy Volunteers taking 600 mg of ACZ885 (Canakinumab) Intravenous (IV) on Day 1.
- ACZ885 (Canakinumab): RA Patients: Patients with Rheumatoid Arthritis RA taking 600 mg of ACZ885 (Canakinumab) Intravenous (IV) on Day 1, Day 15, and Day 43.
Arm/Group | ACZ885 (Canakinumab): Healthy Volunteers | Placebo Comparator: Healthy Volunteers | ACZ885 (Canakinumab): RA Patients | Placebo Comparator: RA Patients
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 2/50 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 4/10 | 12/50 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACZ885 (Canakinumab): Healthy Volunteers (N=10) | Placebo Comparator: Healthy Volunteers (N=10) | ACZ885 (Canakinumab): RA Patients (N=50) | Placebo Comparator: RA Patients (N=10)
Deafness Neurosensory (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Ear Infection (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACZ885 (Canakinumab): Healthy Volunteers (N=10) | Placebo Comparator: Healthy Volunteers (N=10) | ACZ885 (Canakinumab): RA Patients (N=50) | Placebo Comparator: RA Patients (N=10)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 3 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Influenza Like Illness (General disorders) | 1 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 1 | 0
Acute Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory Tract Infection Viral (Infections and infestations) | 0 | 0 | 3 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 1
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 0 | 1
Iron Deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3
Headache (Nervous system disorders) | 2 | 1 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 2 | 1
Phlebitis (Vascular disorders) | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.